CLINICAL TRIAL: NCT01955447
Title: Effect of Different Levels of Plant-based Ingredients on Post-prandial Glucose in Healthy Subjects
Brief Title: Post-prandial Glucose in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: FDS-NAA-1335
Record Dates: First submitted 2013-09-27; First posted 2013-10-07 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2013-11

CONDITIONS: Healthy Subjects
Keywords: Blood glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Reference (Placebo Comparator): no added plant-based ingredients
  Interventions: Dietary Supplement: no added plant-based ingredients to starchy meal
- Low level plant-based ingredients (Active Comparator): Low level addition of plant-based ingredients
  Interventions: Dietary Supplement: Low level plant-based ingredients added to starchy meal
- Medium level plant-based ingredients (Active Comparator): Medium level addition of plant-based ingredients
  Interventions: Dietary Supplement: Medium level plant-based ingredients added to starchy meal
- High level plant-based ingredients (Active Comparator): High level addition of plant-based ingredients
  Interventions: Dietary Supplement: High level plant-based ingredients added to starchy meal

INTERVENTIONS:
Dietary Supplement: no added plant-based ingredients to starchy meal — no added plant-based ingredients to starchy meal
  Arms: Reference
Dietary Supplement: Low level plant-based ingredients added to starchy meal — Low level plant-based ingredients added to starchy meal
  Arms: Low level plant-based ingredients
Dietary Supplement: Medium level plant-based ingredients added to starchy meal — Medium level plant-based ingredients added to starchy meal
  Arms: Medium level plant-based ingredients
Dietary Supplement: High level plant-based ingredients added to starchy meal — High level plant-based ingredients added to starchy meal
  Arms: High level plant-based ingredients

SUMMARY:
The study is designed to determine the extent to which foods containing different levels of plant-based ingredients affect blood glucose responses in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Willing to give consent to participate in the study in writing;
* Healthy male and female subjects, between the age of ≥20 and ≤50 yrs of age at first screening visit;
* Body Mass Index (BMI) between ≥18 and ≤ 25 kg/m2;
* Apparently healthy: no medical conditions which might affect study measurement, as judged by study physician and/or measured by questionnaire, and/or assessed by haematology, blood chemistry and urinalysis;
* Willing to comply to study protocol during the study;
* Agreeing to be informed about medically relevant personal test-results by study physician;
* Willing to refrain from drinking of alcohol on and one day before the blood withdrawal;
* Fasting blood glucose value of volunteer is ≥ 3.4 and ≤ 6.1 mmol/litre (i.e. 62-110 mg/dl) at screening;
* Haemoglobin level within clinically acceptable range (for male 12 to 17 gm/dL and for females 11 to 15 gm / dL; both inclusive) as judged by the research physician.

Exclusion Criteria:

* Being an employee of Unilever or CRO;
* Chronic smokers, tobacco chewers and drinkers;
* Participation in any other biomedical study 3 months before screening visit day of this study and/or participating in any other biomedical study during the screening period;
* Use of medication which interferes with study measurements including vitamins, tonics;
* Reported intense exercise ≥10 h/week;
* Reported weight loss/gain ≥ 10% of body weight in the 6 months preceding screening
* Blood donation for 2 months prior to screening;
* Urine analysis that showed any drug abuse;
* Allergy to any food or cosmetics;
* If female, not being pregnant or planning pregnancy during the study period;
* If female, lactating or has been lactating for 6 weeks before pre-study investigation and/or during the study period.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2013-11; Primary Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Post-prandial blood glucose area under the curve | 120 minutes

SECONDARY OUTCOMES:
Post-prandial insulin area under the curve | 120 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ketul Modi, MBBS, Principal Investigator — Lambda Therapeutics Research Ltd (LTRL)
Locations (1):
- Lambda Therapeutics Research Ltd (LTRL), Ahmedabad, India